CLINICAL TRIAL: NCT01284218
Title: Retrospective Database Study of Real World Abilify Outcomes in Major Depressive Disorder (MDD)
Status: Completed | Type: Observational
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: i3 Innovus (Industry)
Responsible Party: Sponsor
Other Study IDs: CN138-609
Record Dates: First submitted 2011-01-25; First posted 2011-01-26 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Aripiprazole cohort
- Other atypical cohort
- Other antidepressant cohort
- Mood stabilizer cohort
- Stimulant cohort

SUMMARY:
To examine the differences in health care utilization and costs between MDD patients on adjunctive aripiprazole therapy and MDD patients on other augmentation therapies.

ELIGIBILITY:
Inclusion Criteria:

* ≥1 fill for an augmentation therapy medication from Table 1 during the identification period of 01 January 2005 - 30 November 2008.
* 12 months of continuous enrollment with medical and pharmacy benefits each before the index date (pre-index period) and after the index date (post-index period).
* ≥1 medical claim with a primary International Classification of Diseases, 9th Revision, Clinical Modification (ICD-9-CM) diagnosis for MDD (296.2x, 296.3x, 311.xx) during the pre-index period.
* Age ≥18 years as of the year of the pre-index period.

Exclusion Criteria:

* No pharmacy claims for atypical antipsychotics, mood stabilizers, anxiolytics, anticonvulsants, or stimulants, during the pre-index period.
* No medical claims with primary or secondary diagnoses for non-MDD episodic mood disorders or schizophrenia during the pre-index or post-index periods.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Commercial health plan members
Sampling Method: Non-Probability Sample
Enrollment: 23514 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
All cause health care costs | 12 months

SECONDARY OUTCOMES:
Health care costs: MDD related, mental health related | 12 months
Health care resource utilization: All cause, MDD related, mental health related | 12 months
Duration of index therapies | 12 months
Medication possession ratio to evaluate adherence | 12 months
Discontinuation of index therapies | 12 months
Therapy switches to a non-index antidepressant or non-index augmentation therapy | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS Clinical Trials Disclosure — http://www.bms.com/clinical_trials/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: For FDA Safety Alerts and Recalls refer to the following link: http://www.fda.gov/MEDWATCH/safety.htm — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm